CLINICAL TRIAL: NCT06884007
Title: Dikkat Eksikliği ve Hiperaktivite Bozukluğu Olan Çocukların Primer Bakım Verenlerinde Telepsikiyatrik Ebeveyn Eğitimi Programının Etkilerinin İncelenmesi
Brief Title: Effects of Telepsychiatric Parent Training on Caregivers of Children With ADHD (TPT-ADHD)
Acronym: TPT-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 3786-GOA; 2022/3786-GOA (Other: Dokuz Eylul University Ethics Committee)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Telepsychotherapy; Attention Deficit Disorder With Hyperactivity (ADHD); Children; Caregiver; Psychosocial Intervention
Keywords: ADHD; child; caregiver; telepsychiatry; videoconference
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This study employed a parallel-group quasi-experimental design with a pre-test, post-test, and 2-month follow-up. Participants were assigned to either the experimental or control group. The experimental group received a telepsychiatric parent training program consisting of nine 60-minute videoconference sessions, while the control group continued receiving routine treatment and services without additional intervention during the study period. After the study was completed, the control group was also provided with the same training program. Data were collected at three time points: before the intervention, after the intervention, and at the 2-month follow-up. The study aimed to assess the effects of the intervention on caregiving burden, perceived stress, and child behavioral difficulties.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this study, participants were not informed about which group they were assigned to (experimental or control), as this could have influenced their perception and response to the interventions. Participants were randomly assigned to either the experimental or control group by a third-party who was not involved in the study itself. Both the participants and the investigators who interacted with them during the study sessions were blinded to group assignments. Additionally, the outcomes assessor, who evaluated the primary and secondary outcomes, was also blinded to group assignment to ensure objective measurement of the effects of the intervention. This approach aimed to minimize bias and ensure the validity of the results by preventing the influence of prior expectations or knowledge on both participant behavior and data assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telepsychiatric Parent Training Program (Experimental): Participants in this group received Turkey's first "Telepsychiatric Parent Training" program, which consisted of nine 60-minute videoconference sessions aimed at improving caregiver burden, stress, and child behavioral difficulties.
  Interventions: Behavioral: Telepsychiatric Parent Training Program
- Routine Care (Active Comparator): Participants in this group continued with the routine treatment and services provided to caregivers of children with ADHD at the clinic.
  Interventions: Other: Routine Treatment

INTERVENTIONS:
Behavioral: Telepsychiatric Parent Training Program — This study involves a telepsychiatric parent training program for caregivers of children with ADHD. The program includes 9 sessions, each addressing specific topics related to managing ADHD-related behaviors and enhancing parenting strategies. Sessions are primarily delivered through a telepsychiatric platform, such as video conferencing (e.g., Zoom), with additional support provided through text-based communication via platforms like WhatsApp, and, when necessary, follow-up phone calls. The content covers behavior management techniques, stress coping strategies, and skills for managing emotional and behavioral issues in children with ADHD. This intervention is designed to provide accessible, flexible support to caregivers, enhancing their ability to manage their child's condition.
  Arms: Telepsychiatric Parent Training Program
Other: Routine Treatment — Routine treatment and services (no intervention, participants continue with their usual care)
  Arms: Routine Care

SUMMARY:
This study was conducted to examine the effects of a telepsychiatric parent training program implemented for primary caregivers of children with Attention Deficit Hyperactivity Disorder (ADHD).

The study employed a quasi-experimental pre-test, post-test, and re-test control group design. It was conducted from March to June 2022 via videoconferencing with primary caregivers of children aged 7-12 years diagnosed with ADHD, registered at the Child and Adolescent Mental Health Outpatient Clinic of Dokuz Eylül University Hospital. Caregivers in the experimental group completed Turkey's first "Telepsychiatric Parent Training" program, featuring nine 60-minute videoconference sessions. Data were collected using the "Descriptive Information Form," "Zarid Burden Interview (ZBI-22)," "Perceived Stress Scale (PSS-14)," and "Strengths and Difficulties Questionnaire (SDQ)." Data were collected before the program, after the program, and at the 2-month follow-up. The program was also implemented with caregivers in the control group after the research process was completed. Data from the experimental and control groups were analyzed using two-way mixed ANOVA. To determine the effect of the intervention, post-hoc power (β) analysis was conducted using the G*Power 3.1.9.7 program, and the level of statistical significance was set at 0.05. Study hypotheses are:

H1: There is a difference in the average scores of the Caregiving Burden Scale (CBS) for primary caregivers of children with ADHD based on time, group, and the group*time interaction after the application of a parent training program.

H2: There is a difference in the average scores of the Perceived Stress Scale (PSS-14) for primary caregivers of children with ADHD based on time, group, and the group*time interaction after the application of a parent training program.

H3: There is a difference in the average scores of the Strengths and Difficulties Questionnaire (SDQ) for primary caregivers of children with ADHD based on time, group, and the group*time interaction after the application of a parent training program.

All caregivers (100%) successfully completed the program. Caregivers showed significant improvements in caregiving burden, stress levels , and difficulties.

DETAILED DESCRIPTION:
This study explores the effects of a telepsychiatric parent training program designed for primary caregivers of children diagnosed with Attention Deficit Hyperactivity Disorder (ADHD). ADHD is a common neurodevelopmental disorder that significantly impacts children's behavior, attention, and social interactions, leading to challenges for both the children and their caregivers. This study aimed to assess how a structured, remote training program could help caregivers manage these challenges by reducing caregiver burden, stress, and emotional difficulties.

The research employed a quasi-experimental design, involving both experimental and control groups to evaluate the program's effectiveness. The study was conducted from March to June 2022 with caregivers of children aged 7 to 12 years diagnosed with ADHD. Participants were recruited from the Child and Adolescent Mental Health Outpatient Clinic of Dokuz Eylül University Hospital.

Caregivers in the experimental group participated in Turkey's first "Telepsychiatric Parent Training" program, which consisted of nine 60-minute videoconference sessions. The program was delivered remotely, offering flexibility and ease of access for the participants. The training program was specifically designed to provide caregivers with practical tools and strategies for managing the behavioral challenges of children with ADHD. The sessions covered topics such as ADHD symptoms, parenting techniques, emotional regulation, and stress management.

To measure the effectiveness of the program, data were collected at three points: before the program, immediately after the program, and two months following the program. Several established scales were used to assess various aspects of the caregivers' experiences, including the Zarid Burden Interview (ZBI-22) to evaluate caregiving burden, the Perceived Stress Scale (PSS-14) to measure stress levels, and the Strengths and Difficulties Questionnaire (SDQ) to assess emotional and behavioral difficulties in the children. These tools provided a comprehensive view of the impact of the program on both the caregivers and the children.

The data analysis was conducted using two-way mixed ANOVA to assess the differences across time and between the experimental and control groups. The study's findings revealed significant improvements in caregiving burden, stress levels, and child difficulties, with statistical significance observed across pre-test, post-test, and follow-up measurements. These improvements were further supported by post-hoc power analysis, confirming the program's efficacy in addressing the challenges faced by caregivers of children with ADHD.

This study highlights the positive impact of telepsychiatric parent training on reducing stress, caregiving burden, and child difficulties. The success of this program suggests that similar telepsychiatric interventions can be a sustainable and effective model for supporting caregivers, particularly in settings where in-person interventions may be difficult. Additionally, the involvement of psychiatric nurses in delivering such programs may further enhance the effectiveness of the interventions.

Given that this program is the first of its kind in Turkey, it offers valuable insights into the feasibility and effectiveness of telepsychiatric parent training programs. The results support the idea that expanding such programs could provide significant benefits for caregivers, improving their mental health and quality of life while also benefiting the children they care for.

Future studies are recommended to explore the long-term effects of such interventions and assess their feasibility in a broader context, including different populations and settings. Overall, this research contributes to the growing field of telepsychiatry and offers a promising approach for supporting caregivers of children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study.
* Literacy skills (reading and writing ability).
* A primary caregiver of a child diagnosed with ADHD (according to DSM V criteria), aged 7-12 years, currently on medication.
* The primary caregiver must have been responsible for the child's care for at least 3 months.
* The primary caregiver should be 18 years or older.

Exclusion Criteria:

* The child has additional mental health conditions such as intellectual disability, psychotic disorders, post-traumatic stress disorder, bipolar disorder, obsessive-compulsive disorder, or pervasive developmental disorder.
* The caregiver misses more than three sessions of the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Zarit Burden Interview (ZBI-22) | Baseline (pre-test), immediately after the intervention (post-test, approximately Week 9), and follow-up at 2 months post-intervention (approximately Week 17).
  This outcome measures the caregiver burden experienced by parents of children with ADHD. The ZBI-22 assesses various aspects of the emotional, physical, and social burden on caregivers. It evaluates the level of strain experienced by parents in relation to caregiving tasks and their well-being. The total burden score ranges from 0 to 88, with higher scores indicating a greater level of caregiver burden.
  Time Frame: The measurement will be taken at pre-test, post-test, and during a follow-up period after the intervention (i.e., 2 months post-intervention) to assess changes over time and group differences.
Perceived Stress (PSS-14) | Baseline (pre-test), immediately after the intervention (post-test, approximately Week 9), and follow-up at 2 months post-intervention (approximately Week 17).
  This outcome measures the perceived stress levels of caregivers using the PSS-14. The scale assesses the extent to which caregivers feel stress in their daily lives, particularly regarding the challenges of caring for children with ADHD. The total perceived stress score ranges from 0 to 56, with higher scores indicating greater perceived stress.
Emotional and Behavioral Issues in Children (SDQ) | Baseline (pre-test), immediately after the intervention (post-test, approximately Week 9), and follow-up at 2 months post-intervention (approximately Week 17).
  This outcome measures the emotional and behavioral issues in children with ADHD, as reported by their caregivers. The SDQ assesses various domains, including emotional symptoms, conduct problems, hyperactivity/inattention, peer relationships, and prosocial behavior. The total difficulties score ranges from 0 to 40, with higher scores indicating greater emotional and behavioral difficulties.

SECONDARY OUTCOMES:
Time-Related Changes in the Experimental Group | Baseline (Week 0), immediately after the intervention (Week 9), and follow-up at 2 months post-intervention (approximately Week 17).
  This outcome measures the changes in the primary scales (ZBI-22, PSS-14, SDQ) for the experimental group over the course of the study. Specifically, changes between pre-test, post-test, and 2-month follow-up are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Zumra ULKER DORTTEPE, Dr., Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
At this stage, a decision has not yet been made regarding the sharing of individual participant data (IPD) due to the need to review data security procedures to ensure the protection of participants' privacy. Additionally, the research data will be used solely for analysis within the study.

REFERENCES:
- [Background] Dorttepe ZU, Duman ZC. Examination of Telemental Health Practices in Caregivers of Children and Adolescents with Mental Illnesses: A Systematic Review. Issues Ment Health Nurs. 2022 Jul;43(7):625-637. doi: 10.1080/01612840.2021.2013366. Epub 2022 Jan 12. PMID 35021018
- See also: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- Available data/document: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp: https://tez.yok.gov.tr/UlusalT — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp